CLINICAL TRIAL: NCT04048967
Title: Active Learning Norwegian Preschool(er)s
Acronym: ACTNOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Eivind Aadland, Professor, Western Norway University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACTNOW
Record Dates: First submitted 2019-07-16; First posted 2019-08-07 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Preschool Children's Physical Activity, Health and Development
Keywords: Young children; Preschool; Professional development; Physical activity; Physical fitness; Motor skills; Cognition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster randomization of 23 preschools to the intervention group (professional development) and 23 to the control group (standard of care).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Preschool staffs will participate in 50 hours of professional development over 7 months focused on promotion of physical activity in the preschool setting. Staffs and investigators will work together to develop models to ensure children receive 60 minutes per day of moderate-to-vigorous physical activity, 90 minutes per week of motor challenging physical activity, 90 minutes per week of cognitively engaging games/play, and 90 minutes per week of physically active learning.
  Interventions: Behavioral: Professional development
- Control (No Intervention): Staffs receive no professional development and children will receive standard care.

INTERVENTIONS:
Behavioral: Professional development — professional development of preschool staff
  Arms: Intervention

SUMMARY:
Evidence is lacking about scalable, effective and sustainable interventions to increase physical activity and concomitant outcomes in young children. Therefore, the investigators will conduct a large cluster randomized controlled trial investigating the effects of physical activity professional development of preschool staff on preschool physical activity practices and child health and development over 6 and 18 months. The aim is to recruit 60 preschools and 1200 children aged 3-5 years in one county in the western part of Norway to allow for detecting small to moderate effect sizes and ensuring a heterogeneous sample of preschools for the study of implementation. Children's physical development, children's socio-emotional and cognitive development, and intervention implementation will be investigated. The intervention will be developed with strong user involvement from municipalities and relevant stakeholders to facilitate the development of sustainable solutions.

DETAILED DESCRIPTION:
There are growing concerns about low physical activity levels among preschoolers. As 97% of 3-5-year-olds in Norway attend preschool, preschools are unique arenas for intervention, laying the foundation for equitable development of health, human capital, and life opportunities. Yet, evidence of scalable, effective and sustainable interventions to increase physical activity and concomitant outcomes in preschoolers is lacking. Specifically, there is a need to study how the purposeful use of the preschool instructional context can be used to increase moderate-to-vigorous physical activity across a wide range of motor competences to enhance development, cognitively engaging play, and physically active learning. These aspects, in combination, have the potential to simultaneously affect various developmental and learning outcomes, but implementing such a program requires a highly coordinated effort by highly trained individuals. Therefore, the aim of this study is to investigate the effects of an education module, which is designed to result in highly competent preschool staffs having a good understanding of development of motor competence, provision of cognitively engaging play, physically active learning, and pedagogic/didactic approaches and teaching principles to foster physically active and learning preschoolers, on child developmental outcomes. Hopefully, this professional development will promote a physically active lifestyle in the early years that will favorably influence cognition and learning, and provide an efficient, acceptable, and feasible venue to build human capital and provide an early solution to lifelong public health and developmental challenges.

Two main research questions will be tested using both quantitative and qualitative methods, applied to both the child and organizational levels: 1) How does the intervention affect children's physical activity, physical fitness, motor competence, socio-emotional health, self-regulation, executive functions, and learning? 2) How does the intervention interact with different preschool contexts to produce various individual and organizational outcomes?

The proposed research questions will be investigated using a cluster RCT with randomization at the preschool level, including short- (6-month) and long-term (18-month) follow-up. The intervention development will include strong involvement from preschool owners and staff to provide broad support and anchor the project in the preschool sector. Thus, the investigators aim to combine a large-scale experimental study with continuous improvement effort in this sector allowing each preschool's contextual factors to be reflected within the larger cluster RCT. In this model, to make adaptations within each preschool is not considered a lack of fidelity; rather it is a desired process of institutionalization that balances internal and external validity. This balance also overcomes a common criticism of clinical trials as it increases the value for later scaling and dissemination to the real-world settings. In this way, the aim is to create sustainable solutions for improved child development and public health that can be disseminated in the long-term. Thus, the intervention's development, implementation, and evaluation are framed within a "realist RCT" approach. The intervention model is further framed within a socioecological model, placing the preschool as an influential factor for children's health and development. The intervention has two levels; the preschool level and the child level. In response to the challenge of low staff qualifications to implement physical activity, the main component will be a 7-month professional development offered to preschool staff. The intervention is structured as a 15-credit continuing education module that provide staff the opportunity to achieve credits for their efforts. The study is based on the logic model that this professional development will change preschool practices, which will in turn increase and improve children's physical activity opportunities and levels and lead to child developmental effects. Thus, the main aim of the professional development is to provide preschool staff the necessary expertise and resources to intervene on the child level. Researchers will not directly take part in the delivery of the intervention on the child level. The intervention at the child level is derived from hypotheses, theory and evidence relating to the beneficial effects of physical activity on physical, socio-emotional, and cognitive development and have four core components. Central to the ACTNOW intervention is opportunities for children to engage in a variety of meaningful physically active play that brings joy and supports the development of the whole child. By the integration of the four core components, the aim is to provide children opportunities to increase moderate-to-vigorous physical activity across a wide range of motor competencies to enhance development, cognitive engaging play/games, and physically active learning. As such, the core components and dosages promoted are 1) developmentally appropriate moderate-to-vigorous physical activity (60 min/day), 2) motor challenging physical activity (90 min/week), 3) cognitive engaging play/games (90 min/week), and 4) physical activity integrated with learning activities (90 min/week). The intervention will be delivered by the preschool teachers and staff through the use of a wide specter of types of physically active play; from child-initiated and directed free-play at the one end, to adult-initiated child-directed guided play, and adult-directed and initiated structured teacher-led physical activity at the other end.

The study have 2 waves, the first running from August 2019 to June 2021, and the second from August 2020 to June 2022. The professional development provided in Wave 2 will be adjusted based on experiences and findings from Wave 1. Data collection will have 3 main phases; pre-testing performed before randomization, 6-month follow-up performed at the end of the professional development, and 18-month follow-up performed 1 year after completing the professional development. In addition, process evaluation measures will be taken throughout the study.

Derived from a conservative sample size calculation using standard formulas, including correction for the cluster RCT design, it is an aim to recruit a minimum of 60 preschools and 1200 children to the study. This sample size will allow for uncovering statistical significant standardized effect sizes (Cohen's d) of 0.25-0.30.

A range of measures will be taken to examine the interventions effectiveness on a child level (physical activity, physical fitness, motor skills, adiposity, socio-emotional health, self-regulation, executive functions, and learning) and to describe the implementation and adaptation processes taking place in the preschools over 18 months. The realist evaluation includes both quantitative and qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Attending a participating preschool
* Born in 2014, 2015 or 2016 (wave 1) OR 2015, 2016, or 2017 (wave 2)

Exclusion Criteria:

* None

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1265 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Executive function | Change to 18 months
  Inhibition, working memory, and cognitive flexibility by the Early Years Toolbox
Executive function | Change to 6 months
  Inhibition, working memory, and cognitive flexibility by the Early Years Toolbox
Learning | Change to 18 months
  Early math skills and expressive vocabulary by the Early Years Toolbox
Learning | Change to 6 months
  Early math skills and expressive vocabulary by the Early Years Toolbox
Children's socio-emotional health | Change to 18 months
  Child Self-regulation and Behavior Questionnaire (CSBQ), Early Years Toolbox. Includes 33 items rated 1-5 across subscales of cognitive self-regulation, behavioral self-regulation, emotional self-regulation, sociability, prosocial behavior, externalizing problems, and internalizing problems.
Children's socio-emotional health | Change to 6 months
  Child Self-regulation and Behavior Questionnaire (CSBQ), Early Years Toolbox. Includes 33 items rated 1-5 across subscales of cognitive self-regulation, behavioral self-regulation, emotional self-regulation, sociability, prosocial behavior, externalizing problems, and internalizing problems.
Children's self-regulation | Change to 18 months
  Head-Toes-Knees-Shoulders task (HTKS)
Children's self-regulation | Change to 6 months
  Head-Toes-Knees-Shoulders task (HTKS)

SECONDARY OUTCOMES:
Children's physical activity | Change to 18 months
  ActiGraph GT3X+
Children's physical activity | Change to 6 months
  ActiGraph GT3X+
Children's aerobic fitness, muscle strength and power, and speed-agility | Change to 18 months
  PREFIT test battery
Children's aerobic fitness, muscle strength and power, and speed-agility | Change to 6 months
  PREFIT test battery
Children's motor skills | Change to 18 months
  Standardized observation and scoring tool guided by Test of Gross Motor Development-3 and the Preschooler Gross Motor Quality Scale including a total of 9 tasks across locomotor, object control, and balance skills.
Children's motor skills | Change to 6 months
  Standardized observation and scoring tool guided by Test of Gross Motor Development-3 and the Preschooler Gross Motor Quality Scale including a total of 9 tasks across locomotor, object control, and balance skills.
Children's waist circumference | Change to 18 months
  Cm
Children's waist circumference | Change to 6 months
  Cm
Children's body mass index | Change to 18 months
  Calculated from body mass (kg) and height (m); kgm2
Children's body mass index | Change to 6 months
  Calculated from body mass (kg) and height (m); kgm2
Staffs' physical activity | Change to 18 months
  ActiGraph GT3X+
Staffs' physical activity | Change to 6 months
  ActiGraph GT3X+

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Aadland, PhD, Principal Investigator — Western Norway University of Applied Sciences
Locations (1):
- Western Norway University of Applied Sciences, Sogndal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aadland E, Kvalheim OM, Haugland ES, Vabo KB, Aadland KN. Investigating between-group effects of a physical activity intervention across the physical activity intensity spectrum using multivariate pattern analysis. BMC Public Health. 2025 Nov 24;26(1):3. doi: 10.1186/s12889-025-25722-5. PMID 41286789
- [Derived] Aadland KN, Lervag A, Andersen JR, Howard SJ, Ommundsen Y, Aadland E. Effects of a staff physical activity professional development intervention on preschoolers' mental health and self-regulation: The active learning Norwegian Preschool(er)s (ACTNOW) cluster randomised controlled trial. Psychol Sport Exerc. 2024 Nov;75:102705. doi: 10.1016/j.psychsport.2024.102705. Epub 2024 Jul 18. PMID 39029639
- [Derived] Haugland ES, Nilsen AKO, Vabo KB, Pesce C, Bartholomew J, Okely AD, Tjomsland HE, Aadland KN, Aadland E. Effects of a staff-led multicomponent physical activity intervention on preschooler's fundamental motor skills and physical fitness: The ACTNOW cluster-randomized controlled trial. Int J Behav Nutr Phys Act. 2024 Jul 3;21(1):69. doi: 10.1186/s12966-024-01616-4. PMID 38961489
- [Derived] Aadland E, Tjomsland HE, Johannessen K, Nilsen AKO, Resaland GK, Glosvik O, Lykkebo O, Stokke R, Andersen LB, Anderssen SA, Pfeiffer KA, Tomporowski PD, Storksen I, Bartholomew JB, Ommundsen Y, Howard SJ, Okely AD, Aadland KN. Active Learning Norwegian Preschool(er)s (ACTNOW) - Design of a Cluster Randomized Controlled Trial of Staff Professional Development to Promote Physical Activity, Motor Skills, and Cognition in Preschoolers. Front Psychol. 2020 Jul 3;11:1382. doi: 10.3389/fpsyg.2020.01382. eCollection 2020. PMID 32719636
- See also: Project web-page — https://www.hvl.no/en/research/prosjekt/actnow/